CLINICAL TRIAL: NCT05961293
Title: Impact of Peripheral Sensory Stimulation of the Hand in the Treatment of Stroke: A Preliminary Functional MRI Study
Brief Title: NeuroGlove fMRI Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NeuroGlove LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REG-1001
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2023-11

CONDITIONS: Ischemic Stroke, Acute; Stroke
Keywords: Stroke; Ischemic Stroke; Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Cohort (Healthy Cohort) (Other): Healthy participants who participate in 1 study visit. The healthy participant will undergo one functional MRI which using the NeuroGlove.
  Interventions: Device: NeuroGlove
- Treatment Arm (Experimental): The treatment cohort will undergo two functional MRIs once at baseline and the final fMRI will occur six weeks after initial study visit after daily use of the NeuroGlove.
  Interventions: Device: NeuroGlove

INTERVENTIONS:
Device: NeuroGlove — NeuroGlove is a non-invasive device that provides peripheral somatosensory stimulation to the hand of a stroke victim during acute, subacute, or chronic phases of a stroke. NeuroGlove provides sensory stimulation in the forms of pneumatic puffs of air. There is some early evidence that early peripheral sensory stimulation may improve neurological outcomes following an ischemic stroke.

SUMMARY:
This is a prospective, single center, interventional clinical study containing two cohorts the treatment cohort and control cohort. A total of 13 subjects will be enrolled. Three (3) healthy volunteers will be enrolled in the control cohort and undergo imaging only. Ten (10) subjects who have recently experienced a mild to moderate acute ischemic stroke will receive treatment using the NeuroGlove.

DETAILED DESCRIPTION:
This is a prospective, single center, interventional clinical study containing two cohorts the treatment cohort and control cohort. A total of 13 subjects will be enrolled. Three (3) healthy volunteers will be enrolled in the control cohort and undergo imaging only. Ten (10) subjects who have recently experienced a mild to moderate acute ischemic stroke will receive treatment using the NeuroGlove.

Up to 13 subjects enrolled and complete study procedures. There will be 2 cohorts enrolled in the study:

1. Control Cohort: 3 healthy volunteers
2. Treatment Cohort: 10 subjects who have experienced mild to moderate stroke symptoms* that did not completely resolve after acute interventions.

   * Mild to moderate stroke symptoms is defined as a NIHSSS score of 3 to 15.

ELIGIBILITY:
Inclusion Criteria (control cohort):

* Able and willing to provide informed consent.
* Men and women ≥18 and <85 years of age.
* Subject must be right hand dominant.
* Subject should not have any physical limitations of either upper extremity (e.g., fracture, joint deformity, severe spasticity/contracture, wounds, skin breakdown, lymphedema, etc.)

Inclusion Criteria (treatment cohort):

* Able to and willing to provide informed consent. Legally authorized representatives (LARs) will not be allowed to consent on behalf of the subject.
* Men and women ≥18 and <85 years of age.
* First single acute ischemic stroke with an onset date within 14 days (± 7 days from onset) of enrollment (time of informed consent) into the study.
* Mild to moderate acute ischemic stroke defined as NIHSS score of 3 to 15.
* Measurable weakness of one upper extremity without complete paralysis (detectable movement in at least 3 fingers).
* Subject must be right hand dominant.

Exclusion Criteria:

* Coma, inability to cooperate with the study based on impaired level of consciousness or confusion.
* Known neurological deficit prior to stroke (including but not limited to previous stroke, MS, Parkinson's disease).
* Physical limitations of the weak upper extremity (e.g., fracture, joint deformity, severe spasticity/contracture, wounds, skin breakdown, lymphedema, etc.)
* Any contraindication to the imaging required per the protocol.
* Complete middle cerebral artery infarction based on imaging.
* Carotid artery stenosis >50% of the normal diameter segment (diameter stenosis, compared to the angiographically normal proximal or distal segment).
* Subjects has a known history of substance abuse (drug) or alcohol dependence, or lacks the ability to comprehend or following instructions, or for any reason, in the opinion of the investigator, would be unlikely or unable to comply with study protocol requirements.
* If female, subject is pregnant at the time of enrollment or planning to become pregnant during the trial period.
* Subject has any other acute or chronic condition that the investigator believes will adversely affect the ability to interpret the data or will prevent the subject from completing the trial procedures.
* Currently participating in another interventional clinical trial. (Observational clinical trial participation is allowed for study enrollment.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Brian Function | 6 weeks
  Evaluate brain function through a fMRI assessing post-stroke changes in brain activation including functional recruitment of new brain territories in subjects undergoing rehabilitation with the NeuroGlove.
Rate of Adverse Events | 6 weeks
  Rate and severity of adverse events related to the use of the NeuroGlove.

SECONDARY OUTCOMES:
Motor Recovery | 6 weeks
  Evaluate the motor recovery of the affected upper extremity based on the change in hand grip strength from baseline using hand dynamometer
NIHSS score | 6 weeks
  Evaluate neurological recovery as measure by the change in the National Institutes of Health Stroke Scale (NIHSS) score from baseline. The lower the score less severe the stroke symptoms.
Rankin Score | 6 weeks
  Evaluate functional recovery as measured by the modified Rankin Scale (mRS) score. A 0-6 scale is used to measure degree of ability 0 is no disability and 6 is death.
Change in QOL | 6 weeks
  Change in stroke-specific quality of life (SS-QOL) scores from baseline. Scale is 49-245 with higher scores indicating better function.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Nussbaum, Principal Investigator — NeuroGlove LLC

IPD SHARING:
Plan to Share IPD: No
There is no plan for sharing individual participants data to other researchers.